CLINICAL TRIAL: NCT00154063
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel-Group Study to Evaluate the Efficacy and Safety of E2007 in Migraine Prophylaxis
Brief Title: Efficacy and Safety Study of E2007 in Migraine Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-A001-210; NCT00239941 (obsolete NCT alias)
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2009-08

CONDITIONS: Migraine Prophylaxis
MeSH Terms: interventions — perampanel

ARMS (2):
- Placebo (Placebo Comparator): During the Titration Phase, placebo was initiated at a dose of 1.0 mg/day for the first 2 weeks, increased to 1.5 mg/day for the next 2 weeks, and then further increased to 2.0 mg/day for 10 weeks (last 2 weeks of the Titration Phase continuing into the 8-week Maintenance Phase).
  Interventions: Other: Placebo
- E2007 (Experimental): During the Titration Phase, perampanel was initiated at a dose of 1.0 mg/day for the first 2 weeks, increased to 1.5 mg/day for the next 2 weeks, and then further increased to 2.0 mg/day for 10 weeks (last 2 weeks of the Titration Phase continuing into the 8-week Maintenance Phase).
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007
  Arms: E2007
Other: Placebo
  Arms: Placebo

SUMMARY:
This was a 22-week, prospective, randomized, double-blind, placebo-controlled, multicenter, parallel-group study that included a 4-week Baseline Phase at the beginning and a 4-week single-blind placebo Safety Phase at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any race, 18 to 65 years of age inclusive.
2. Patients with a history of migraine (with or without aura) according to the Headache Classification Committee of the IHS. Migraine attacks have to have had an onset before age 50 and have to have been present for at least 12 months.
3. Patients with 4-12 qualified migraine attacks per month over the past three months prior to Screening, as well as during the four weeks of the Baseline Phase will be eligible for entry into this study. The interval between two qualified migraine attacks should be at least 24 hours to be counted as distinct migraine attacks. A qualified migraine attack without aura is defined as a headache that lasts 4-72 hours (if untreated or unsuccessfully treated) or if successfully treated (revised per Amendment 01). This attack has at least two of the following characteristics: unilateral location, pulsating quality, moderate or severe intensity that inhibits or prohibits daily activities or aggravation by routine physical activities such as walking up stairs. In addition, at least one of the following symptoms must be present during the headache: nausea, vomiting, or photophobia and phonophobia (revised per Amendments 01 and 02). A qualified migraine attack with aura must fulfill the same criteria as the headache attack, plus have an associated aura as defined by the Migraine Criteria of the Headache Classification Committee of the International Headache Society. An aura alone that requires acute migraine treatment will also be considered a migraine attack.
4. Male and female patients will be eligible for enrollment. Females should be either of non-childbearing potential by reason of surgery, radiation, menopause (one year post onset), or of childbearing potential and practicing a medically acceptable method of contraception (eg, abstinence, a barrier method plus spermicide, or IUD) for at least one month before study randomization and for two months after the end of the study, and have a negative serum B-hCG at Screening. Pregnant and/or lactating females are excluded. Those women using hormonal contraceptives must also be using an additional approved method of contraception (eg, a barrier method plus spermicide, or IUD) starting with the Baseline Phase and continuing throughout the entire study period.
5. Patients with a Body Mass Index (BMI) between 19 to 40 kg/m2 inclusive at Screening.
6. Patients who are willing to participate and have provided written informed consent prior to being exposed to any study-related procedures.

Exclusion Criteria:

1. Patients with chronic daily headaches as defined by more than 14 headache days per month on average during the three months prior to Screening,
2. Patients with cluster headaches and other trigeminal autonomic cephalalgias, and other primary headaches (except tension-type headache) and secondary headaches (defined according to the Headache Classification Committee of the IHS 2004),
3. Patients with a history of being non-responsive to more than two classes of adequately conducted, prophylactic migraine treatments (e.g., beta blockers, calcium channel blockers, tricyclics, MAOIs, valproate (divalproex), topiramate, gabapentin),
4. Patients who use the following medications as described:

   * Use of marketed triptans for 10 days or greater per month on average,
   * Use of ergot-containing medications for ten days or greater per month on average,
   * Use of NSAIDs, acetaminophen, or isometheptene-containing agents for 15 days or greater per month on average,
   * Use of opioids for 10 days or greater per month on average,
   * Use of any two or more of the above medications for 15 days or greater per month on average,
5. Patients with clinically significant neurological illness, other than migraine, that, in the opinion of the Investigators, may have the potential of altering pain perception or reporting,
6. Patients with a history of or currently having major psychiatric disorders including schizophrenia, major depressive disorder, or bipolar disorder,
7. Patients who are known to be positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV),
8. Patients with elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) >= 1.5 times the upper limit of normal (ULN),
9. Patients with evidence of significant active hematological disease; white blood cell count cannot be less than or equal to 2500/uL or an absolute neutrophil count less than or equal to 1000/uL,
10. Patients with clinically significant ECG abnormality, including prolonged QTc (Fridericia correction) defined as >= 450 msec for males and >= 470 msec for females,
11. Patients with clinically significant active hepatic disease, cardiovascular, metabolic, respiratory, renal, endocrinological, gastrointestinal diseases, and bacterial or viral infections within 30 days prior to Screening or during the Baseline Phase,
12. Patients with known or suspected history of alcoholism or drug abuse within the previous two years, or a positive finding on urinary drug screening of other than prescribed medications,
13. Patients who have had severe allergic reactions to multiple drugs,
14. Patients with any other condition that would make them, in the opinion of the PI, unsuitable for this study,
15. Patients that have participated in a study involving administration of an investigational compound (including E2007) within one month of Visit 1 (Screening),
16. Patients with a known or suspected allergy to lactose, excluding lactose intolerance,
17. Patients who use the following medications for any medical reason during the study: beta-blockers, tricyclic antidepressants, antiepileptics, calcium channel blockers, monoamine oxidase inhibitors, NSAIDs daily, magnesium supplements at high doses (ie, 600 mg/day), riboflavin at high doses (ie, 100 mg/day), corticosteroids, local anesthetics, botuliunum toxin, or herbal preparations such as feverfew or St. John's Wort. Patients who use non-pharmacological prophylactic approaches that were started at least one month prior to Screening may be continued throughout the study.
18. (revised per Amendment 03)
19. Patients who fail to complete the migraine diary adequately during the Baseline Phase (ie, patients, who do not have complete diary entries for at least 21 days of the Baseline Phase).

Randomized patients will be both male and female, 18-65 years of age, of any race, with a history of migraine headaches (with or without aura according to the Headache Classification Committee of the International Headache Society (IHS, 2004 guideline) for at least 12 months, with an onset before age 50, experiencing 4-12 migraine attacks per month during both the 3 months prior to Screening and the Baseline Phase. Patients' Body Mass Index (BMI) should be between 19 to 40 kg/m2 inclusive at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Young, M.D., Ph.D., Study Director — Eisai Inc.
Locations (9):
- United States (9):
  - Investigational Site, Oceanside, California
  - Investigational Site, Santa Monica, California
  - Investigational Site, Tampa, Florida
  - Investigational Site, West Palm Beach, Florida
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Springfield, Missouri
  - Elkind Headache Center, Mount Vernon, New York
  - Investigational Site, Greensboro, North Carolina
  - Investigational Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | E2007
Started | 104 | 102
Completed | 92 | 80
Not Completed | 12 | 22
Not completed — Adverse Event | 4 | 8
Not completed — Protocol Violation | 1 | 1
Not completed — Investigator or Sponsor Request | 0 | 1
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | E2007 | Total
Number analyzed (Participants) | 104 | 102 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (11.5) | 41.3 (12.5) | 41.4 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Male and female (either of non-childbearing potential, childbearing potential and practicing a medically acceptable method of contraception, surgically sterile, or postmenopausal for greater or equal to 1 year) subjects with a history of migraine experiencing 4 to 12 migraine attacks per month during both the 3 months prior to Screening and the Baseline Phase.
  Participants
    Female | 90 | 89 | 179
    Male | 14 | 13 | 27

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Average Duration Per Migraine Attack in Treatment Phase (LOCF)
Description: The duration of a migraine attack was the sum of the duration (in hours) of each migraine headache that was collapsed to form the migraine attack. The time between the offset of first migraine headache and the onset of the next migraine headache was not counted in the duration of migraine attack. The average duration of the migraine attacks in each phase was calculated as the total duration (in hours) of the migraine attacks during each phase, divided by the number of migraine attacks in the corresponding treatment phase. Efficacy analyses were performed using both the 24-hour and 48-hour rule. The data is presented as mean hours +/- standard error.
Time Frame: Baseline to Week 19
Population: ITT Population
Measure: Mean (Standard Error); unit: Hours
Groups:
- Placebo (24 Hour Rule); Placebo (48 Hour Rule): During the Titration Phase, placebo was initiated at a dose of 1.0 mg/day for the first 2 weeks, increased to 1.5 mg/day for the next 2 weeks, and then further increased to 2.0 mg/day for 10 weeks (last 2 weeks of the Titration Phase continuing into the 8-week Maintenance Phase).
- E2007 (24 Hour Rule); E2007 (48 Hour Rule): During the Titration Phase, perampanel was initiated at a dose of 1.0 mg/day for the first 2 weeks, increased to 1.5 mg/day for the next 2 weeks, and then further increased to 2.0 mg/day for 10 weeks (last 2 weeks of the Titration Phase continuing into the 8-week Maintenance Phase).
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Hours | 0.69 (1.79) | 4.65 (3.27) | -1.22 (2.16) | 3.70 (3.58)

2. Secondary Outcome: Change From Baseline in Average Migraine Severity Per Migraine Attack in Treatment Phase (LOCF)
Description: The average migraine attack severity in each treatment phase was calculated using the sum of the severity of migraine attacks during the treatment phase, divided by the number of qualified migraine attacks. The scale of severity for each migraine attack ranges from 0 to 100, with higher scores indicating increased migraine severity. Efficacy analyses were performed using both the 24-hour and 48-hour rule.
Time Frame: Baseline to Week 19
Population: ITT Population
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Units on a Scale | 0.95 (1.23) | 0.26 (1.09) | 0.97 (1.22) | 0.19 (1.09)

3. Secondary Outcome: Change From Baseline in Migraine Attack Frequency Per 28 Days in Treatment Phase (LOCF)
Description: Qualified migraine headache was defined as two major subtypes: migraine without aura(headache that lasted 4-72 hours with at least two characteristics: unilateral location, pulsating quality, moderate/ severe pain intensity or aggravation by/ causing avoidance of routine physical activity and either nausea/ vomiting or photophobia,phonophobia); migraine with aura (attack with reversible focal neurological symptoms that usually precede or sometimes accompany the headache) per Migraine Criteria of the Headache Classification Committee of the International Headache Society. All of the qualified headaches, which occur after the initial qualified migraine headache, but within 24 hours of previous qualified migraine headache, were collapsed into one qualified migraine attack. Two qualified migraine attacks were considered to be distinct when the end of previous and the beginning of the next migraine attack were separated by at least 24/48 hours per 24/48 hour rule.
Time Frame: Baseline to Week 19
Population: ITT Population
Measure: Mean (Standard Error); unit: Migraine attack
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Migraine attack | -2.06 (0.20) | -1.95 (0.24) | -1.51 (0.15) | -1.49 (0.20)

4. Secondary Outcome: Change From Baseline in Migraine Period Frequency Per 28 Days in Maintenance Phase
Description: A migraine period was defined as a migraine headache that started, ended, or recurred within 24 hours. If the headache persisted for longer than 24 hours, it was considered a new migraine period. Efficacy analyses were performed using both the 24-hour and 48-hour rule for defining migraine periods. Data is presented as mean number of migraine period per 28 days +/- standard error. A negative change indicates a decrease in the number of migraine periods from baseline.
Time Frame: Baseline, Week 11 to Week 19
Population: ITT Population
Measure: Mean (Standard Error); unit: Migraine period
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Migraine period | -2.9 (0.35) | -2.91 (0.38) | -3.27 (0.40) | -3.52 (0.43)

5. Primary Outcome: Change From Baseline in Migraine Period Frequency Per 28 Days in Treatment Phase (LOCF)
Description: A migraine period was defined as a migraine headache that started, ended, or recurred within 24 hours. If the headache persisted for longer than 24 hours, it was considered a new migraine period. Participants recorded the frequency of migraine period in diary. Efficacy analyses were performed using both the 24-hour and 48-hour rule for defining migraine periods. Data is presented as mean number of migraine period per 28 days +/- standard error. A negative change indicates a decrease in the number of migraine periods from baseline. LOCF = last observation carried forward (ie, observation from last phase with active treatment)
Time Frame: Baseline to Week 19
Population: The efficacy analysis was performed on the Intention to treat (ITT) Population, which was defined as all randomized subjects who received at least 1 dose of double-blind study medication, and had baseline and postbaseline migraine assessments in at least 1 phase.
Measure: Mean (Standard Error); unit: Migraine period
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Migraine period | -2.94 (0.32) | -2.73 (0.39) | -3.31 (0.39) | -3.00 (0.50)

6. Secondary Outcome: Change From Baseline in Number of Days Requiring Symptomatic Rescue Medication Per 28 Days in Treatment Phase (LOCF)
Description: The number of days requiring symptomatic rescue medication was calculated as the number of calender days during the migraine attack when the patient took one or more migraine rescue medications as recorded on the participant's diary. The calendar date(s) during which medication was taken will be used for calculations. Efficacy analyses were performed using both the 24-hour and 48-hour rule. The data is presented as mean days +/- standard error.
Time Frame: Baseline to Week 19
Population: ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Days | -3.05 (0.38) | -2.74 (0.44) | -3.10 (0.38) | -2.68 (0.48)

7. Secondary Outcome: Change From Baseline in Number of Days With Migraine Attack Per 28 Days in Treatment Phase (LOCF)
Description: A migraine attack day was defined as a calendar day (from 0 hours to 24 hours) during which at least one migraine attack took place. If the migraine attack continues through midnight, each day will be counted separately. Efficacy analyses were performed using both the 24-hour and 48-hour rule. Data is presented as mean number of days with migraine attack per 28 days +/- standard error.
Time Frame: Baseline to Week 19
Population: ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Days | -3.77 (0.39) | -3.27 (0.47) | -4.1 (0.43) | -3.48 (0.56)

8. Secondary Outcome: Change From Baseline in Number of Participants With Patient Global Impression of Change (PGIC) of Migraine (LOCF)
Description: The PGIC was a self-evaluation scale for each patient to assess his or her status compared to baseline in migraine headache frequency and intensity, the occurrence of adverse events, and overall functional status, measured on a 7-point scale. The scale ranges from "very much improved" with a score of 1 to "very much worse" with a score of 7. A responder is defined as being "very much improved" or "much improved". The data is presented as number of participants. LOCF = last observation carried forward (ie, observation from last phase with active treatment)
Time Frame: Baseline to Week 23
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 104 | 101
Participants
  Very Much/Much Improved | 40 | 41
  No Change/Minimally Improved | 56 | 52
  Worsened | 8 | 8

9. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Headache Pain Score
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 7, pain due to headache was assessed on a scale of 0-10 with 0 being no pain and 10 being the most painful.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 95 | 90
units on a scale | -0.83 (2) | -0.28 (2)

10. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Headaches
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 6, the number of days with headache (Headache which lasted more than one day was counted as each day) was assessed. The data is presented as mean days +/- standard deviation.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 95 | 91
Days | -6.80 (13) | -6.99 (11)

11. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Less Housework
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 4, the number of days when productivity in household work reduced by half of more because of a headache was assessed. The data is presented as mean days +/- standard deviation.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 95 | 91
Days | -3.4 (8) | -2.3 (7)

12. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Less Work or School
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 2, the number of days with reduced productivity by at least half at school or work because of a headache was assessed. The data is presented as mean days +/- standard deviation.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 94 | 90
Days | -1.76 (7) | -2.47 (7)

13. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Missed Housework
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 3, the number of days when participant skipped performing household chores or regular household activities because of a headache was assessed. The data is presented as mean days +/- standard deviation.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 94 | 91
Days | -3.07 (7) | -2.45 (7)

14. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Missed Non-Work Activities
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 5, the number of days when participant miss leisure or social activities because of a headache was assessed. The data is presented as mean days +/- standard deviation.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 95 | 91
Days | -1.34 (4) | -2.07 (6)

15. Secondary Outcome: Change From Baseline of Migraine Disability Assessment Questionnaire Score (MIDAS) at Week 23: Missed Work or School
Description: The MIDAS questionnaire was a participant assessed 7-item questionnaire designed to measure the impact of headache in the last 3 months. Based on question 1 , the number of missed work or school because of a headache was assessed. The data is presented as mean days +/- standard deviation.
Time Frame: Baseline, Week 23
Population: ITT Population. Only patients with non-missing baseline data are summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | E2007
Number analyzed (Participants) | 94 | 90
Days | -1.20 (3) | -0.82 (3)

16. Secondary Outcome: Percentage of Participants With a Greater Than or Equal to 50% Decrease in Migraine Attack Frequency Per 28 Days in Treatment Phase (LOCF)
Description: as for outcome 3
Time Frame: Week 5 to Week 19
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Percentage of Participants | 46.2 | 47.5 | 36.5 | 45.5

17. Secondary Outcome: Percentage of Participants With a Greater Than or Equal to 50% Decrease in Migraine Period Frequency Per 28 Days in Treatment Phase (LOCF)
Description: A migraine period was defined as a migraine headache that started, ended, or recurred within 24 hours. If the headache persisted for longer than 24 hours, it was considered a new migraine period. Participants recorded the frequency of migraine period in diary. Efficacy analyses were performed using both the 24-hour and 48-hour rule for defining migraine periods. The data is presented as percentage of participants.
Time Frame: Week 5 to Week 19
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo (24 Hour Rule) | E2007 (24 Hour Rule) | Placebo (48 Hour Rule) | E2007 (48 Hour Rule)
Number analyzed (Participants) | 104 | 101 | 104 | 101
Percentage of Participants | 48.1 | 50.5 | 51.9 | 52.5

ADVERSE EVENTS:
Time Frame: From baseline (day 1) up to 30 days after participant's treatment end date or final study visit or up to week 23.
Description: Treatment emergent adverse events (TEAEs), defined as an AE that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication are presented in this section. The data presented in the other AE section includes serious adverse events.
Arm/Group | Placebo | E2007
Serious Adverse Events (participants affected / at risk) | 1/104 | 1/102
Other Adverse Events (participants affected / at risk) | 75/104 | 74/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | E2007 (N=102)
Abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | E2007 (N=102)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 2
Eye pain (Eye disorders) | 2 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Toothache (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1
?Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 7 | 6
Influenza like illness (General disorders) | 2 | 1
Pain (General disorders) | 1 | 2
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 1
Feeling cold (General disorders) | 1 | 1
Malaise (General disorders) | 2 | 0
Thirst (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Injected limb mobility decreased (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Injection site swelling (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pre-existing condition improved (General disorders) | 0 | 1
Sluggishness (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Tenderness (General disorders) | 0 | 1
Liver tenderness (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Multiple allergies (Immune system disorders) | 0 | 1
?Seasonal allergy (Immune system disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 14 | 10
Upper respiratory tract infection (Infections and infestations) | 9 | 11
Urinary tract infection (Infections and infestations) | 8 | 6
Sinusitis (Infections and infestations) | 5 | 6
Fungal infection (Infections and infestations) | 4 | 3
Gastroenteritis viral (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 5 | 2
Bronchitis (Infections and infestations) | 4 | 1
Streptococcal infection (Infections and infestations) | 4 | 0
Viral infection (Infections and infestations) | 0 | 3
Herpes zoster (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Dental caries (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Vaginal candidiasis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3
Joint sprain (Injury, poisoning and procedural complications) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
?Back injury (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Human bite (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 4
Protein urine present (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Bacteria urine (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood urine present (Investigations) | 1 | 1
Crystal urine present (Investigations) | 1 | 1
White blood cells urine positive (Investigations) | 1 | 1
Blood potassium abnormal (Investigations) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Cardiac murmur functional (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Gastric pH decreased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haematology test abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Mean cell volume decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 1 | 0
Urinary sediment present (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 9 | 10
Somnolence (Nervous system disorders) | 4 | 7
Migraine (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 4 | 1
Sinus headache (Nervous system disorders) | 2 | 3
Sedation (Nervous system disorders) | 1 | 3
Lethargy (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 2 | 0
Ageusia (Nervous system disorders) | 1 | 0
Anosmia (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
?Mental impairment (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Nightmare (Psychiatric disorders) | 1 | 1
Aggression (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Thinking abnormal (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
?Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Onychorrhexis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Hot flush (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No